CLINICAL TRIAL: NCT00003205
Title: A Phase II Trial of Bryostatin-1 for the Treatment of Stage IV Breast Cancer
Brief Title: Bryostatin 1 in Treating Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 97-0751.cc; UCHSC-97751; NCI-T97-0063
Record Dates: First submitted 1999-11-01; First posted 2003-04-23 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2002-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — bryostatin 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of bryostatin 1 in treating patients with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical response of patients with stage IV breast cancer to bryostatin 1.
* Determine the efficacy of this regimen in these patients.
* Estimate the pharmacokinetic parameters of bryostatin 1 when given as 24 hour infusion.
* Determine the ability of this regimen to regulate lymphocyte function in these patients.
* Determine the effect of this regimen on platelet function and protein kinase C activity in these patients.

OUTLINE: Patients receive bryostatin 1 IV over 24 hours. Treatment continues weekly in the absence of disease progression or unacceptable toxicity.

Patients are followed every 4-8 weeks for tumor response.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Unequivocal diagnosis of metastatic breast cancer
* Bidimensionally measurable disease
* No uncontrolled CNS metastases
* No disease that is evaluable only, including blastic bone disease, malignant ascites, and malignant pleural effusion
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Menopausal status:

* Not specified

Performance status:

* SWOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* At least 18 weeks

Hematopoietic:

* Platelet count at least 50,000/mm^3
* PT and PTT within normal limits
* Neutrophil count at least 2,000/mm^3

Hepatic:

* Bilirubin no greater than 1.2 mg/dL
* Transaminases no greater than 3 times normal

Renal:

* Creatinine no greater than 1.6 mg/dL OR
* Creatinine clearance at least 70 mL/min

Other:

* No active infections requiring antibiotics
* No viral hepatitis allowed
* Seronegative for hepatitis B or C
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 2 months following study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* 2 prior chemotherapy regimens for metastatic disease allowed as adjuvant therapy or for advanced disease (may include high dose chemotherapy with stem cell support)
* At least 4 weeks since prior chemotherapy
* At least 6 weeks since prior nitrosourea or mitomycin therapy
* No other concurrent chemotherapy

Endocrine therapy:

* 2 prior hormonal therapy regimens for metastatic disease as adjuvant therapy or for advanced diseases allowed
* At least 2 weeks since prior hormonal therapy (at least 4 weeks in case of disease progression while receiving hormonal therapy after initial response)
* No concurrent hormonal therapy except oral contraceptives
* No concurrent use of steroids except for management of severe or life- threatening toxic effects arising from bryostatin 1

Radiotherapy:

* At least 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No concurrent use of drugs known to interfere with platelet function, such as aspirin or NSAIDs (including ibuprofen)
* No concurrent use of anticoagulants
* At least 2 weeks since prior use of aspirin
* At least 2 days since prior use of NSAIDS
* Concurrent use of acetaminophen to control pain is allowed
* If acetaminophen inadequate for pain control, concurrent use of oral narcotics such as codeine or oxycodone is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Kraft, MD, Study Chair — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Denver, Colorado, United States